CLINICAL TRIAL: NCT02320903
Title: Phase I - Using Mobile Technology to Enhance MST Outcomes (VillageWhere)
Brief Title: Using Mobile Technology to Enhance Multisystemic Therapy (MST) Outcomes
Acronym: VillageWhere
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Evidence-Based Practice Institute, Seattle, WA (Industry)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1R43MH097349-01 (NIH); 1R43MH097349-01 (NIH)
Record Dates: First submitted 2014-12-16; First posted 2014-12-19 (Estimated); Results first posted 2018-02-14 (Actual); Last update posted 2018-02-14 (Actual); Status verified 2017-11

CONDITIONS: Child Behavior Disorders
Keywords: Criminal Justice; Juvenile Delinquency
MeSH Terms: conditions — Child Behavior Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Use of VillageWhere App Prototype (Experimental): In this single-arm study design, all enrolled caregivers and teens will use the VillageWhere App Prototype that has been developed for this study. They are requested to use it as often as they would like throughout the duration of the trial. The app is designed to be used several times throughout each day.
  Interventions: Device: VillageWhere App

INTERVENTIONS:
Device: VillageWhere App

SUMMARY:
The goal of the current trial is to assess the feasibility of a newly developed prototype of a cell phone app called VillageWhere. VillageWhere is designed to improve clinical outcomes of youth with externalizing behavioral problems by improving parental monitoring of youth whereabouts and activities while increasing the delivery of rewards to teens for good behavior. This Phase I Small Business Innovation Research (SBIR) proposal seeks to develop and conduct initial feasibility testing of the VillageWhere prototype. The primary features of the prototype include location monitoring via smartphones' global positioning system (GPS) functionality as well as facilitating teen self-appraisal of meeting behavioral expectations. Good behavior is rewarded with points that are tracked by the app and can be used to redeem for real-world rewards. The investigators will conduct an 45-day open trial (N=20 caregiver/teen dyads) to assess use, feasibility and acceptability for teens involved in the juvenile justice system or otherwise struggling with externalizing behavioral problems. Caregivers and teens will be assessed at baseline, before receiving the app, and at the end of the app use period (45 days). The therapist of each caregiver/teen dyad will also be assessed at the end of the app use period. Primary outcomes include: use of app features, monitoring of teen behavior and whereabouts, delivery of real-world rewards, and feasibility and acceptability. Secondary outcomes include: parenting behaviors, externalizing teen behaviors and internalizing teen behaviors.

DETAILED DESCRIPTION:
VillageWhere was pilot tested with a sample of 16 youth and their primary caregiver participating in an EST for a serious conduct problem (Mean age 14.6 years, 52% male, 56% African American, 33% were previously arrested). After completing baseline self-report measures, dyads used the app as desired for 4 weeks, then participated in a post-assessment and qualitative interviews. App usage by both parents and youth was high with little diminished use over the four weeks of the trial. All parents set and used reinforcers for functional behavior and used the "find my teen" feature; 84% set geolocation expectations for youth's whereabouts at specific times; and 88% set other expectations for the youth (e.g., finish homework), viewed notifications, and regularly used the "Find My Teen" feature. As expected, parents interacted with the app frequently: 2.4 times per day. Youth used the app on average four times per day. All youth earned and redeemed points for complying with their parent's expectations and routinely viewed their behavior plans (93.3%) and feedback notification messages (86.7%). Parents did not on average use coaching videos (20%).

Although the study was not powered to detect statistical significance, a series of paired t-tests were conducted to examine pre- to post-changes on self-report measures. Changes for parents and youth all were in predicted directions, with effect sizes ranging from small to high (average d = .42, range .21-.80). Parents reported greater use of positive parenting behaviors (i.e., rewards and praise), greater discipline consistency, lower overall perceived stress, a higher feeling of influence over youth behavior, and greater parenting efficacy. Youth reported increases in parent use of positive behaviors, consistency, and knowledge of whereabouts. Parent- and youth-reported change in youth aggression and rule-breaking (as measured by the CBCL/YSR).

Qualitative results were also positive. Using 7-point scales, parents and youth reported on app satisfaction three times/week. Parent ratings were high (M = 6.0) across items (e.g., "The app was helpful today," "I have ways to intervene with my teen"). Youth satisfaction scores were also high (M = 6.1; e.g., "My parent is noticing & rewarding my good behavior;" "I liked getting app prompts & reminders"). Parents reported that the app helped them trust their youth, increase their use of rewards, and made giving rewards easier; they also reported a reduction in youths' "excuse-making." Youth perceived that the app allowed them more freedom, because parents had an objective way of verifying their whereabouts. Nearly all youth (89%) liked that their parent was more consistent in paying attention to their positive behaviors and rewarding them for it (versus only being punitive). Both parents and youth described significant improvements in their relationship.

In addition, 16 therapists working with the parent-youth dyads also gave qualitative feedback that was highly positive. Therapists stated that they liked the extra accountability the app afforded to teens and the reduction in parent-youth communication issues.

ELIGIBILITY:
Inclusion Criteria:

* Teen: English speaking, between ages of 13 and 17, juvenile justice involvement and/or externalizing behavioral problems, currently in treatment and will remain in treatment for duration of trial
* Caregiver: English speaking, owns Android smart phone, currently in treatment with their teen and will remain in treatment for duration of trial

Exclusion Criteria:

* N/A

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2014-04; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda A. Dimeff, PhD, Principal Investigator — Evidence-Based Practice Institute; Cindy M Schaeffer, PhD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- Evidence-Based Practice Institute, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We completed a four-week within-subjects pre-post trial to determine the usability, acceptability, and feasibility. MST therapists in Seattle, New York City, Hartford, and Washington, DC referred families to the study. Parents contacted the study team to indicate their interest. Therapists of referred families also were enrolled in the study.
Pre-assignment Details: Initial App Set Up: Clinicians were solely responsible for assisting families to set up their app; however, many clinicians were uncomfortable with this because they were not "tech savvy". Solution: Phase II will include a self-guided setup tool that will empower users (parents, youth) to complete the set up independently.
Groups:
- Therapists; Parents/Caregivers; Youth/Teens: In this study, all enrolled caregivers and teens will be referred to the study by their participating therapists. All caregiver/teen dyads will use the VillageWhere App Prototype that has been developed for this study. They are requested to use it as often as they would like throughout the duration of the trial. The app is designed to be used several times throughout each day.
  VillageWhere App
Period: Overall Study
Arm/Group | Therapists | Parents/Caregivers | Youth/Teens
Started | 24 | 32 | 32
Completed | 16 | 16 | 16
Not Completed | 8 | 16 | 16
Not completed — Withdrawal by Subject | 0 | 9 | 9
Not completed — Exited therapy; no longer eligible | 8 | 2 | 2
Not completed — Lost to Follow-up | 0 | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Therapists | Parents/Caregivers | Youth/Teens | Total
Number analyzed (Participants) | 24 | 32 | 32 | 88
Age, Continuous [Mean (Standard Deviation); unit: Years] — Demographics collected only for parents and teens who completed the study (parents=16, teens=16) Population: Demographics reported only for families that completed the study.
  Years
    Age: number analyzed (Participants) | 0 | 16 | 16 | 32
    Age |  | 41.7 (0) | 14.6 (1.6) | 24.15 (0)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Demographics reported only for families that completed the study.
  Participants
    number analyzed (Participants) | 24 | 16 | 16 | 56
    Female | 22 | 15 | 9 | 46
    Male | 2 | 1 | 7 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 3 | 8
  Not Hispanic or Latino | 20 | 12 | 11 | 43
  Unknown or Not Reported | 2 | 17 | 18 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 5 | 5 | 11
  White | 5 | 9 | 8 | 22
  More than one race | 0 | 1 | 1 | 2
  Unknown or Not Reported | 17 | 17 | 18 | 52
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24 | 32 | 32 | 88

OUTCOME MEASURES:

1. Primary Outcome: App Usage - Parent Set up / Modified an App-based Behavior Plan for the Teen
Description: Percent of parents who set up a behavior plan for teen using app features.
Time Frame: up to 45-days
Population: All parent/caregiver and teen participants analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- Parents/Caregivers: All caregivers who used the VillageWhere App Prototype that was developed for this study. They were requested to use it as often as they would like throughout the duration of the trial. The app is designed to be used several times throughout each day.
  VillageWhere App
Arm/Group | Parents/Caregivers
Number analyzed (Participants) | 16
Participants | 16

2. Primary Outcome: App Usage - Set up and Allocated / Earned Points (Rewards) for Positive Teen Behavior
Description: How many parents/caregivers set up a reward system and redeemed at least some points for the teen.
Time Frame: up to 45-days
Population: Percent of caregivers who set and allocated points to the teen (teens who had points redeemed).
Measure: Count of Participants; unit: Participants
Groups:
- Parents/Caregivers: All caregiver/teen dyads used the VillageWhere App Prototype that was developed for this study. They were requested to use it as often as they would like throughout the duration of the trial. The app is designed to be used several times throughout each day.
  VillageWhere App
Arm/Group | Parents/Caregivers
Number analyzed (Participants) | 16
Participants | 16

3. Primary Outcome: App Usage - Parent Set Geolocation Expectations for the Teen.
Description: Percentage of parent/caregivers who set either required or off-limits locations for their teens.
Time Frame: up to 45-days
Measure: Count of Participants; unit: Participants
Groups:
- Parents/Caregivers: In this single-arm study design, all enrolled caregivers and teens will use the VillageWhere App Prototype that has been developed for this study. They are requested to use it as often as they would like throughout the duration of the trial. The app is designed to be used several times throughout each day.
  VillageWhere App
Arm/Group | Parents/Caregivers
Number analyzed (Participants) | 16
Participants | 14

4. Primary Outcome: App Usage - Viewed Notifications Regarding Behavioral Expectations Met/Not Met
Description: The percentage of participants who viewed notifications that the teen was or was not meeting a behavioral expectation. Both parents and teens had this capability.
Time Frame: up to 45 days
Population: All parent/caregiver and teen participants analyzed
Measure: Count of Participants; unit: Participants
Groups:
- Youth/Teens: All caregiver/teen dyads used the VillageWhere App Prototype that was developed for this study. They were requested to use it as often as they would like throughout the duration of the trial. The app is designed to be used several times throughout each day.
  VillageWhere App
Arm/Group | Parents/Caregivers | Youth/Teens
Number analyzed (Participants) | 16 | 16
Participants | 14 | 14

5. Primary Outcome: App Usage - Viewed Parent Coaching Videos
Description: The app included 5 brief video vignettes depicting an effective parenting technique.
Time Frame: up to 45 days
Population: Only the parent/caregiver version of the app had this feature.
Measure: Count of Participants; unit: Participants
Groups:
- Parents/Caregivers Only: Parent/caregiver users of the linked parent-youth phone app system.
Arm/Group | Parents/Caregivers Only
Number analyzed (Participants) | 16
Participants | 3

6. Primary Outcome: App Usage - View Progress Graph (Points Earned Over Time)
Description: Youth/teen points earned over time were depicted on a graph for each day of use. To view the graph, caregivers/parents and youth/teens had to click on an app button.
Time Frame: up to 45 days
Population: Analyses performed separately for parents and teens.
Measure: Count of Participants; unit: Participants
Arm/Group | Parents/Caregivers | Youth/Teens
Number analyzed (Participants) | 16 | 16
Participants | 10 | 8

7. Primary Outcome: App Satisfaction Rating - the App Was Helpful Today
Description: Parent/caregiver was prompted randomly 3 times each week to rate on a scale of 1 (strongly disagree) to 7 (completely agree), how helpful was the app to you today?
Time Frame: up to 45 days
Population: Only parent/caregivers were administered this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Parents/Caregivers
Number analyzed (Participants) | 16
units on a scale | 5.95 (.999)

8. Primary Outcome: App Satisfaction Rating - I Have Ways to Intervene With my Teen.
Description: Parent/caregiver was prompted randomly 3 times each week to rate on a scale of 1 (strongly disagree) to 7 (completely agree), the app gives me new ways of intervening with my teen.
Time Frame: up to 45 days
Population: Only parent/caregivers were given this question.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Parents/Caregivers Only
Number analyzed (Participants) | 16
units on a scale | 6.00 (1.09)

9. Primary Outcome: App Satisfaction Rating - Overall Satisfaction
Description: Parent/caregiver and teen was prompted randomly 3 times each week to rate on a scale of 1 (totally unsatisfied) to 7 (completely satisfied), overall, how satisfied are you with the app today?
Time Frame: up to 45 days
Population: Parent/caregiver and teen participants were analyzed separately on this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Parents/Caregivers | Youth/Teens
Number analyzed (Participants) | 16 | 16
units on a scale | 5.91 (1.21) | 6.14 (0.72)

10. Primary Outcome: App Satisfaction Rating - Parent is Noticing and Rewarding Good Behavior
Description: Three times each week, at random, youth/teens were asked to rate on a scale of 1 (strongly disagree) to 7 (strongly agree), my parent is noticing and rewarding good behavior. All ratings were averaged across full period of app use.
Time Frame: up to 45 days
Population: Only youth/teens were provided this question.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Youth/Teens Only: Youth/teens who used the app.
Arm/Group | Youth/Teens Only
Number analyzed (Participants) | 16
units on a scale | 6.19 (1.15)

11. Primary Outcome: App Satisfaction - I Like Getting Prompts and Reminders
Description: Youth/teens in the study were prompted 3 times/week during period of app usage to rate, on a scale of 1 (strongly disagree) to 7 (strongly agree), "I like getting prompts and reminders from the app."
Time Frame: up to 45 days
Population: Only teens were provided with this question.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Youth/Teens Only
Number analyzed (Participants) | 16
units on a scale | 5.62 (1.27)

12. Secondary Outcome: Achenbach System of Empirically-Based Assessment, Aggression Subscale
Description: The Achenbach System of Empirically-Based Assessment is a measure of youth problem behavior and psychiatric symptomatology that has parallel parent (report of teen) and youth (self-report) versions to allow for different perspectives on the problem. The parent version is called the Child Behavior Checklist (CBCL) and the youth version is called the Youth Self Report (YSR). Selected subscales from the CBCL and the YSR were administered before and after the 4 weeks of app usage, in this case, the aggression subscale. Higher values indicate worse symptoms. Possible range on this subcale is 0 - 36; a score of 13 or higher indicates clinically significant aggression, defined as aggression that is higher than that of 93% of teens in the United States.
Time Frame: Baseline and Post assessment (end of 45-day app use period)
Population: Parent/caregivers and youth/teens results were analyzed separately.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Parents/Caregivers | Youth/Teens
Number analyzed (Participants) | 16 | 16
units on a scale
  Mean at Time 1 (baseline) | 13.75 (8.80) | 11.29 (4.82)
  Mean at Time 2 (post-usage) | 12.31 (8.80) | 10.14 (5.43)
Statistical Analysis 1: Comparison: Parents/Caregivers; Paired sample T tests were used to measure change for parents over time; Test type: Equivalence — What was the within-group change over time effect size (Cohen's d)?; Paired samples T test (change over time); Cohen's d for parent report on this measure was 0.16
Statistical Analysis 2: Comparison: Youth/Teens; Paired sample T tests were used to measure change over time for teens; Test type: Equivalence — What was the within-group change over time effect size (Cohen's d)?; Paired samples T test (change over time); Cohen's d for youth report was d = 0.22

13. Secondary Outcome: Achenbach System of Empirically-Based Assessment, Depression Subscale
Description: The Achenbach System of Empirically-Based Assessment is a measure of youth problem behavior and psychiatric symptomatology that has parallel parent (report of teen) and youth (self-report) versions to allow for different perspectives on the problem. The parent version is called the Child Behavior Checklist (CBCL) and the youth version is called the Youth Self Report (YSR). Selected subscales from the CBCL and the YSR were administered before and after the 4 weeks of app usage, in this case, the depression subscale. Higher values indicate worse symptoms. Possible range on this subcale is 0 - 26; a score of 8 or higher indicates clinically significant depression, defined as depressive symptoms higher than that of 93% of teens in the United States.
Time Frame: Baseline and Post assessment (end of 45-day app use period)
Population: Parent/caregivers and youth/teens results were analyzed separately. Least squares means show amount of difference from pre- to post-testing in paired samples T tests.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Parents/Caregivers | Youth/Teens
Number analyzed (Participants) | 16 | 16
units on a scale
  Pre-test mean | 6.93 (5.36) | 6.29 (4.81)
  Post-test mean | 5.80 (5.17) | 4.71 (3.91)
Statistical Analysis 1: Comparison: Parents/Caregivers; Paired sample T tests were used to measure change for parents over time; Test type: Equivalence — What was the within-group change over time effect size (Cohen's d)?; Paired samples T test (change over time); Cohen's d for parent report on this measure was d = 0.22
Statistical Analysis 2: Comparison: Youth/Teens; Paired sample T tests were used to measure change for teens over time; Test type: Other — What was the within-group change over time effect size?; Cohen's d for teen report on this measure was d = 0.22

14. Secondary Outcome: Achenbach System of Empirically-Based Assessment, Rule-breaking Subscale
Description: The Achenbach System of Empirically-Based Assessment is a measure of youth problem behavior and psychiatric symptomatology that has parallel parent (report of teen) and youth (self-report) versions to allow for different perspectives on the problem. The parent version is called the Child Behavior Checklist (CBCL) and the youth version is called the Youth Self Report (YSR). Selected subscales from the CBCL and the YSR were administered before and after the 4 weeks of app usage, in this case, the rule-breaking subscale. Higher values indicate worse symptoms. Possible range on this subcale is 0 - 34; a score of 9 or higher indicates clinically significant rule-breaking, defined as rule-breaking that is higher than that of 93% of teens in the United States.
Time Frame: Baseline and Post assessment (end of 45-day app use period)
Population: Parent/caregivers and youth/teens results were analyzed separately.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Parents/Caregivers | Youth/Teens
Number analyzed (Participants) | 16 | 16
units on a scale
  Mean at Time 1 (baseline) | 9.71 (6.34) | 10.07 (4.20)
  Mean at Time 2 (post-usage) | 9.07 (6.49) | 9.21 (4.61)
Statistical Analysis 1: Comparison: Parents/Caregivers; Paired sample T tests were used to measure change for parents over time; Test type: Equivalence — What was the within-group change over time effect size (Cohen's d)?; Paired samples T test (change over time); Cohen's d for parent report on this measure was d = 0.10
Statistical Analysis 2: Comparison: Youth/Teens; Paired samples T tests were used to measure change over time for teens; Test type: Equivalence — What was the within-group change over time effect size? (Cohen's d); Cohen's d for youth report was d = 0.28

15. Secondary Outcome: Loeber Parental Supervision Scale
Description: This measure of extent to which parents supervise and monitor youth whereabouts was administered to parents/caregivers and to youth/teens before and after the 4 weeks of app usage.This 8-item scale has a scored range of 0 (minimum score) - 16 (maximum score), with high scores indicating more or better parental supervision/monitoring.
Time Frame: Baseline and Post assessment (end of 45-day app use period)
Population: Parent/caregivers and youth/teens results were analyzed separately.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Parents/Caregivers | Youth/Teens
Number analyzed (Participants) | 16 | 16
units on a scale
  Mean at Time 1 (baseline) | 13.00 (2.25) | 10.86 (3.32)
  Mean at Time 2 (post-usage) | 13.38 (2.45) | 11.50 (2.44)
Statistical Analysis 1: Comparison: Parents/Caregivers; Paired sample T tests were used to measure change for parents over time; Test type: Equivalence — What was the within-group change over time effect size (Cohen's d)?; Paired samples T test (change over time); Cohen's d for parent report on this measure was d = 0.16
Statistical Analysis 2: Comparison: Youth/Teens; Paired sample T tests were used to measure change for teens over time; Test type: Equivalence — What was the within-group change over time effect size? (Cohen's d); Cohen's d for youth report was d = 0.21

16. Secondary Outcome: Loeber Positive Parenting Scale
Description: This measure of extent to which parents express warmth and encouragement to youth was administered to parents/caregivers and to youth/teens before and after the 4 weeks of app usage.This 9-item scale has a scored range of 0 (minimum score) - 18 (maximum score), with high scores indicating more parental positivity.
Time Frame: Baseline and Post assessment (end of 45-day app use period)
Population: Parent/caregivers and youth/teens results were analyzed separately.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Parents/Caregivers | Youth/Teens
Number analyzed (Participants) | 16 | 16
units on a scale
  Mean at Time 1 (baseline) | 8.87 (4.97) | 8.57 (2.24)
  Mean at Time 2 (post-usage) | 11.39 (2.95) | 8.93 (2.79)
Statistical Analysis 1: Comparison: Parents/Caregivers; Paired sample T tests were used to measure change for parents over time; Test type: Equivalence — What was the within-group change over time effect size (Cohen's d)?; Paired samples T test (change over time); Cohen's d for parent report on this measure was d = 0.62
Statistical Analysis 2: Comparison: Youth/Teens; Paired sample T tests were used to measure change over time for teens; Test type: Equivalence — What was the within-group change over time effect size (Cohen's d)?; Cohen's d for youth report was d = 0.23

17. Secondary Outcome: Loeber Parental Consistency Scale
Description: This measure of extent to which parents are consistent in their rules, expectations, and discipline techniques with youth was administered to parents/caregivers and to youth/teens before and after the 4 weeks of app usage. This 5-item scale has a scored range of 0 (minimum score) - 10 (maximum score), with high scores indicating more consistent / better parental discipline follow-through.
Time Frame: Baseline and Post assessment (end of 45-day app use period)
Population: Parent/caregivers and youth/teens results were analyzed separately.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Parents/Caregivers | Youth/Teens
Number analyzed (Participants) | 16 | 16
units on a scale
  Mean at Time 1 (baseline) | 1.87 (1.64) | 5.21 (2.01)
  Mean at Time 2 (post-usage) | 2.27 (2.02) | 5.57 (2.87)
Statistical Analysis 1: Comparison: Parents/Caregivers; Paired sample T tests were used to measure change for parents over time; Test type: Equivalence — What was the within-group change over time effect size (Cohen's d)?; Cohen's d for parent report on this measure was d = 0.22
Statistical Analysis 2: Comparison: Youth/Teens; Paired samples T tests were used to measure within-groups change over time for teens; Test type: Equivalence — What was the within-group change over time effect size (Cohen's d)?; Cohen's d for youth report was d = 0.26

18. Secondary Outcome: Loeber Parental Effectiveness Scale
Description: Degree to which parents feel that their parenting techniques are working in terms of managing teen behavior challenges. This 3-item scale has a scored range of 0 (minimum score) - 8 (maximum score), with high scores indicating better discipline effectiveness (e.g., "I feel like the punishment I give works in curbing youth behavior").
Time Frame: Change over 30 days of app usage (baseline to post-assessment)
Population: All parents/caregivers who completed the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Parents/Caregivers Only
Number analyzed (Participants) | 16
units on a scale
  Mean at Time 1 (baseline) | 4.20 (1.90)
  Mean at Time 2 (post-usage) | 4.40 (1.88)
Statistical Analysis 1: Comparison: Parents/Caregivers Only; Paired sample T tests were used to measure change for parents over time; Test type: Equivalence — What was the within-group change over time effect size (Cohen's d)?; Cohen's d for parent report on this measure was d =.12

19. Secondary Outcome: Perceived Stress Scale (PSS)
Description: Degree to which parents are experiencing stress related to parenting. This 10-item scale has a scored range of 0 (minimum score) - 40 (maximum score), with high scores indicating more stress related to parenting.
Time Frame: Change over 30 days of app usage (baseline to post-assessment)
Population: All parents/caregivers who completed the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Parents/Caregivers Only
Number analyzed (Participants) | 16
units on a scale
  Mean at Time 1 (baseline) | 18.09 (8.14)
  Mean at Time 2 (post-usage) | 12.73 (4.45)
Statistical Analysis 1: Comparison: Parents/Caregivers Only; Paired sample T tests were used to measure change for parents over time; Test type: Equivalence — What was the within-group change over time effect size (Cohen's d)?; Cohen's d for parent report on this measure was d = 0.81

20. Secondary Outcome: Parental Locus of Control Scale
Description: Degree to which parents feel efficacious and confident in managing parenting challenges. This 20-item scale has a scored range of 0 (minimum score) - 40 (maximum score), with high scores indicating that the parent has a higher sense of feeling efficacious in their role as a parent.
Time Frame: Change over 30 days of app usage (baseline to post-assessment)
Population: All parents/caregivers who completed the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Parents/Caregivers Only
Number analyzed (Participants) | 16
units on a scale
  Mean at Time 1 (baseline) | 15.25 (6.22)
  Mean at Time 2 (post-usage) | 18.63 (8.72)
Statistical Analysis 1: Comparison: Parents/Caregivers Only; Paired sample T tests were used to measure change for parents over time; Test type: Equivalence — What was the within-group change over time effect size (Cohen's d)?; Cohen's d for parent report on this measure was d = 0.43

21. Secondary Outcome: Loeber Parental Knowledge Scale
Description: Youth report of how much parents actually know about the youth's whereabouts/activities. This 5-item scale has a scored range of 0 (minimum score) - 15 (maximum score), with high scores indicating that the parent knows more about what teens are actually doing.
Time Frame: over 30 days of app usage
Population: Youth/teens who used app only
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Youth/Teens Only
Number analyzed (Participants) | 16
units on a scale
  Mean at Time 1 (baseline) | 8.07 (2.73)
  Mean at Time 2 (post-usage) | 9.00 (3.09)
Statistical Analysis 1: Comparison: Youth/Teens Only; Paired sample T tests were used to measure change for teens over time; Test type: Equivalence — What was the within-group change over time effect size (Cohen's d)?; Cohen's d for youth report on this measure was d = 24

ADVERSE EVENTS:
Time Frame: Adverse events were informally monitored throughout the 4-week period during which time parents and teens were using the app. Also, most families had their baseline assessment sessions 1-2 weeks prior to the start of app use, and their post-assessment 1-2 weeks after finishing their use of the app. Thus, adverse events were informally monitored for the entire study period, for most families, approximately 8 weeks.
Description: Since the study was non-medical, participants were NOT at risk of a mortality event, i.e., the intervention involved use of a phone app only. Participants were also not at risk for a serious adverse event involving "a life-threatening event, hospitalization, or incapacity/disability." As a social science study, our participants may have had some risk of Other including Not Serious Adverse events, such as embarrassment or discomfort answering psychologically- and behaviorally-oriented questions.
Groups:
- Use of VillageWhere App Prototype: In this single-arm study design, all enrolled caregivers and teens used the VillageWhere App Prototype that was developed for this study. They were requested to use it as often as they would like throughout the duration of the trial. The app is designed to be used several times throughout each day. Thus, the risk was identical for both parents and teens, since both experienced the app as the only intervention (i.e., there was no comparison group who did not use the app).
Arm/Group | Use of VillageWhere App Prototype
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-09-12): https://cdn.clinicaltrials.gov/large-docs/03/NCT02320903/Prot_SAP_000.pdf